CLINICAL TRIAL: NCT06339541
Title: La Piattaforma ACC di Ricerca Preclinica Per l'Oncologia di Precisione
Brief Title: The ACC Preclinical Research Platform for Precision Oncology
Acronym: ACC Platform
Status: Recruiting | Type: Observational
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Collaborators: Alleanza Contro il Cancro (Other)
Responsible Party: Principal Investigator, Enzo Medico, Head of Oncogenomics, Fondazione del Piemonte per l'Oncologia
Other Study IDs: 029-FPO23
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor; Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Solid and haematological tumor tissues, blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ACC Preclinical Research Platform for Precision Oncology is a retrospective and prospective observational study focused on the implementation and validation of the application of PDCM (Patient Derived Cancer Models) generated from tissues or cells of patients with neoplastic disease, as a tool to improve molecular and biological knowledge of tumours and to test the efficacy and sensitivity of pharmacological treatments.

DETAILED DESCRIPTION:
This is a retrospective and prospective observational study, focused on the implementation and validation of the application of PDCM, generated from tissue or cells of patients, including paediatric patients, with solid and haematological malignancies, as a tool to improve molecular and biological knowledge of tumours and to test the efficacy and sensitivity of pharmacological treatments.

An up-to-date database of all PDCMs available at the participating italian hospitals will be generated and enriched with new models generated during the course of the project. The sharing of models and procedures between the different hospitals will facilitate their molecular and phenotypic characterisation, also in parallel with the tumours of origin, as well as their validation as tools for testing the efficacy of drugs for precision medicine. By establishing common workflows and standards and performing cross-validation experiments it is planned to build a network of reference centres as a resource for drug screening on 2D and 3D models.

ELIGIBILITY:
Inclusion Criteria:

* Patients, including paediatric patients, with solid and haematological malignancies for whom tissue or tumour cell material is available.

Exclusion Criteria:

* none

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, including paediatric patients, with solid and haematological malignancies for whom tissue or tumour cell material is available.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
number of PDCM (patient derived cancer models) | 12 months
  PDCM will be generated from tissues and cells
number of Whole Exome Sequencing (WES) e RNA-seq performed | 12 months
  WES and RNA seq will be performed on tissues and blood

SECONDARY OUTCOMES:
number of PDCM shared within the network | 12 months
  PDCM will be generated from tissues and cells and shared within the network

CONTACTS AND LOCATIONS:
Overall Officials: Enzo Medico, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia
Locations (1):
- Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo, Candiolo, Turin, Italy